CLINICAL TRIAL: NCT06626685
Title: Clonal Hematopoiesis of Indeterminate Potential in Heart Failure - RICO-HF.
Brief Title: Clonal Hematopoiesis of Indeterminate Potential in Heart Failure.
Acronym: RICO-HF
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: RICO-HF
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study of clonal hematopoiesis requires the use of sequencing technologies, as the Next Generation Sequencing (NGS), currently employed in the diagnosis and therapy of solid tumors and hematological malignancies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Heart Failure: Patients hospitalized with acute HF classified according to LVEF.
  Interventions: Other: Clinical and instrumental examination
- Chronic Heart Failure: Ambulatory patients with chronic HF classified according to LVEF.
  Interventions: Other: Clinical and instrumental examination

INTERVENTIONS:
Other: Clinical and instrumental examination — Each patient, consecutively afferent to the SC Cardiologia I of the ASST-PG23 in Bergamo with the diagnosis of acute or chronic HF, at enrollment will undergo to routine clinical and instrumental examination.

SUMMARY:
This study is part of the Rico Macro-Project, a multidisciplinary research program promoted by FROM in collaboration with the ASST-PG23 and ATS Bergamo, aiming to investigate the role of clonal hematopoiesis on inflammation, studying in depth the mechanisms underlying the inflammatory process to determine their correlation with some important pathologies in different clinical fields (Hematology, Cardiology, Neurology, Pneumology, Gastroenterology, and Diabetology, etc.). In this context, the prospective observational study RICO-HF is developed.

The RICO HF is the first project focused on CHIP and inflammation in the area of Cardiology, specifically in HF.

DETAILED DESCRIPTION:
CHIP is associated with a pro-inflammatory state and its mechanistic link to HF has been demonstrated in animal and cellular models, and in patient cohorts (14-24).

Although HF in humans has various causes, different pathophysiological mechanisms and heterogeneous clinical manifestations, the experimental and clinical data reported so far support the relevance of inflammatory cytokine production and signaling by immune cells in the pathogenesis of cardiac dysfunction and HF.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients admitted to the Cardiology Unit of the ASST Papa Giovanni XXIII Hospital, Bergamo for acute HF and patients attending the outpatient HF clinic of the same hospital for chronic HF
* age >18 years
* written informed consent

Exclusion Criteria:

* chronic therapy with anti-inflammatories, steroids, immunomodulators, immunosuppressants, chemotherapeuthic agents
* previous heart transplant
* cardiogenic shock or cardiac arrest
* recent acute coronary syndrome (<3 months)
* current acute infection requiring specific treatment
* overt MPNs
* primary myelodysplastic syndromes
* malignant cancers
* non-cardiovascular co-morbidity reducing life expectancy to < 1 year
* any factor precluding 1-year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consecutively afferent to the SC Cardiologia I of the ASST-PG23 Hospital in Bergamo with the diagnosis of acute or chronic Heart Failure.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the prevalence of CHIP in patients with a diagnosis of acute HF according to the value of LVEF>50% (HFpEF) or ≤50% (HFmrEF/HFrEF) at the time of hospitalization. | At diagnosis during the baseline
  Obtained by medical health records

SECONDARY OUTCOMES:
Estimation of CHIP prevalence in patients with acute HFpEF, by de novo and worsening conditions | At baseline; 1 year follow-up.
  Obtained by medical health records
Estimation of CHIP prevalence in HF patients, according to the acute or chronic conditions and classified by LVEF | At baseline; 1 year follow-up.
  Obtained by medical health records
Association between CHIP and patterns of inflammatory biomarkers in patients with acute de novo HFpEF | At baseline; 1 year follow-up.
  Obtained by medical health records
Association between CHIP and outcome (mortality, urgent heart transplant, HF hospitalization and need for urgent visit due to HF decompensation) | At baseline; 1 year follow-up.
  Obtained by medical health records
Association between CHIP and patients' clinical characteristics at baseline | At baseline; 1 year follow-up.
  Obtained by medical health records

CONTACTS AND LOCATIONS:
Overall Officials: ANTONELLO GAVAZZI, MD, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (2):
- Italy (2):
  - ATS BERGAMO Agenzia di Tutela della Salute, Bergamo
  - Asst Papa Giovanni Xxiii - Dip. Di Cardiologia, Bergamo